CLINICAL TRIAL: NCT01053000
Title: Photodynamic Therapy With Levulan® Topical Solution And Blue Light +/- Topical Retinoid Pre-Treatment In The Treatment Of Dorsal Hand/Forearm Actinic Keratoses
Brief Title: Photodynamic Therapy With Levulan® +/- Topical Retinoid Pre-Treatment In The Treatment Of Actinic Keratoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stewart, Roger H., M.D., P.A. (Other)
Responsible Party: Principal Investigator, Barry Galitzer, MD, Physician, Stewart, Roger H., M.D., P.A.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INV-0901
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Results first posted 2015-07-22 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-07

CONDITIONS: ACTINIC KERATOSES
Keywords: ACTINIC KERATOSES; HAND; FOREARM
MeSH Terms: conditions — Keratosis, Actinic | interventions — tazarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lt. Arm Tazorac/Rt. Arm No Pretreatment (Experimental): Apply Tazorac 0.1% gel for 1 week to the Left arm only and then receive ALA- PDT Treatment to both arms
  Interventions: Drug: Tazorac
- Rt. Arm Tazorac/Lt. Arm No Pretreatment (Experimental): Apply Tazorac 0.1% gel for 1 week to the Right arm only and then receive ALA- PDT Treatment to both arms
  Interventions: Drug: Tazorac

INTERVENTIONS:
Drug: Tazorac — compare the safety and efficacy of broad area photodynamic therapy with aminolevulinic acid (ALA-PDT) following topical retinoid pre-treatment with Tazorac vs ALA-PDT with occlusion only (no pretreatment) in subjects with dorsal hand/forearm actinic keratoses, with an incubation time of 60 minutes, using blue light.
  Other Names: tazarotene

SUMMARY:
To determine and compare the safety and efficacy of broad area photodynamic therapy with aminolevulinic acid (ALA-PDT) following topical retinoid pre-treatment vs ALA-PDT with occlusion only (no pretreatment) in subjects with dorsal hand/forearm actinic keratoses, with an incubation time of 60 minutes, using blue light.

DETAILED DESCRIPTION:
Subjects will be randomized such that their RIGHT dorsal hand/forearm will receive one of the following two treatments with the subject's LEFT dorsal hand/forearm receiving the other treatment; Treatment 1 will include pre-treatment of the dorsal hand/forearm with Tazorac 0.1% gel BID for one week, followed by ALA applied to the entire dorsal hand/forearm 60 minutes prior to BLUE light treatment for 16 minutes 40 seconds Treatment 2 will have ALA applied to the entire dorsal hand/forearm and occluded for 60 minutes prior to BLUE light treatment for 16 minutes 40 secondsNote: ALA will be applied to individual dorsal hand/forearm actinic keratoses (AK) lesions followed by broad area application over the entire dorsal hand/forearm surface. The treatment area on the side NOT pre-treated with Tazorac will then be occluded using plastic wrap for 60 minutes. The treatment area of the dorsal hand/forearm is defined as the extensor surface of the hand/forearm between the elbow and the base of the fingers (the fingers are NOT included in the treatment area).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or non-pregnant female over the age of 18 years. Females must be post-menopausal, surgically sterile or using a medically acceptable form of birth control, with a negative urine pregnancy test at the Baseline visit. 2. Subject has provided written and verbal informed consent.

3. Subject has at least four (4) AK lesions (Grade 1 or 2) on each Treatment Area (dorsal forearm/hand surface), with at least 3 of these lesions in a continuous 25 cm2 Target Area on the hand or forearm.

4. Subject is willing to comply with study instructions and return to the clinic for required visits.

Exclusion Criteria:

* 1. Subject is pregnant, lactating, or is planning to become pregnant during the study.

  2. Subject has a history of cutaneous photosensitization, porphyria, hypersensitivity to porphyrins or photodermatosis or any condition with associated immunosuppression (e.g. HIV, systemic malignancy, etc.).

  3. Subject has any skin pathology or condition that could interfere with the evaluation of the test product or requires the use of interfering topical or systemic therapy.

  4. Subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.

  5. Subject is currently enrolled in an investigational drug or device study. 6. Subject has received an investigational drug or been treated with an investigational device within 30 days prior to the initiation of treatment (baseline).

  7. Subject is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.

  8. Subject may be unreliable for the study including subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits.

  9. Subject has a known sensitivity to one or more of the vehicle components (ethyl alcohol, isopropyl alcohol, laureth 4, polyethylene glycol).

  10. Subject has a known sensitivity to one or more of the components of Tazorac (tazarotene, benzyl alcohol, ascorbin acid, butylated hydroxyanisole, butylated hydroxytoluene, carbomer 934P, edentate disodium, hexylene glycol, poloxamer 407, polyethylene glycol 400, polysorbate 40, tromethamine).

  11. Subject has the need to be exposed to artificial tanning devices or excessive sunlight during the trial.

  12. Subject has used photosensitizing drugs, (e.g. thiazides, tetracyclines, fluoroquinolones, phenothiazines, sulfonamides, etc) within a timeframe where photosensitization from these drugs may still be present, or has the need to use them during the trial.

  13. Subject has used any of the following topical preparations on the dorsal hands/forearms:· Keratolytics including urea (greater than 5%), alpha hydroxyacids [e.g. glycolic acid, lactic acid, etc. greater than 5%], salicylic acid (greater than 2%) within 2 days of initiation of treatment. · Retinoids, including tazarotene, adapalene, tretinoin, retinol, within 4 weeks of the initiation of treatment.· 5-FU, cryotherapy, diclofenac, imiquimod or other treatments for AK within 8 weeks of initiation of treatment.· Microdermabrasion, laser ablative treatments or chemical peels within 8 weeks of the initiation of treatment. · ALA-PDT within 6 months of initiation of treatment.

  14. Subject has used any of the following systemic medications: · Immuno-suppressants including steroids, chemotherapy, etc. within 3 months of the initiation of treatment· Retinoid therapy within 6 months of the initiation of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Galitzer, MD, Principal Investigator — Roger H. Stewart MD PA
Locations (1):
- Roger Stewart MD PA, Fort Lauderdale, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Left Arm Tazorac/Right Arm No Tazorac Pre-treatment: Tazorac 0.1% gel was applied for 1 week to the left arm followed by therapy with aminolevulinic acid (ALA-PDT) to both arms, in subjects with dorsal hand/forearm actinic keratoses, with an incubation time of 60 minutes, using blue light.
- Right Arm Tazorac/Left Arm No Pretreatment: Tazorac 0.1% gel was applied for 1 week to the right arm followed by therapy with aminolevulinic acid (ALA-PDT) to both arms, in subjects with dorsal hand/forearm actinic keratoses, with an incubation time of 60 minutes, using blue light.
Period: Overall Study
Arm/Group | Left Arm Tazorac/Right Arm No Tazorac Pre-treatment | Right Arm Tazorac/Left Arm No Pretreatment
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Tazorac o.1% gel foer 1 week to the randomly chosen arm
  20% aminolevulinic acid HCL: compare the safety and efficacy of broad area photodynamic therapy with aminolevulinic acid (ALA-PDT) following topical retinoid pre-treatment vs ALA-PDT with occlusion only (no pretreatment) in subjects with dorsal hand/forearm actinic keratoses, with an incubation time of 60 minutes, using blue light.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Lesion Counts in 25 cm2 Target Area Relative to Baseline.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- Tazorac Treated Arm: Tazorac o.1% gel for 1 week to the randomly chosen arm
  20% aminolevulinic acid HCL: compare the safety and efficacy of broad area photodynamic therapy with aminolevulinic acid (ALA-PDT) following topical retinoid pre-treatment in subjects with dorsal hand/forearm actinic keratoses, with an incubation time of 60 minutes, using blue light.
- No Pretreatment With Tzorac: No pretreatmnet to the randomly chosen arm
  20% aminolevulinic acid HCL: compare the safety and efficacy of broad area photodynamic therapy with aminolevulinic acid (ALA-PDT) only (no pretreatment) in subjects with dorsal hand/forearm actinic keratoses, with an incubation time of 60 minutes, using blue light.
Arm/Group | Tazorac Treated Arm | No Pretreatment With Tzorac
Number analyzed (Participants) | 10 | 10
lesions | -72 (30.3) | -37.5 (41.7)

ADVERSE EVENTS:
Groups:
- No Pretreatment Arm: No Pretreatment to the randomly chosen arm
  20% aminolevulinic acid HCL: compare the safety and efficacy of broad area photodynamic therapy with aminolevulinic acid (ALA-PDT) with occlusion only (no pretreatment) in subjects with dorsal hand/forearm actinic keratoses, with an incubation time of 60 minutes, using blue light.
Arm/Group | Tazorac Treated Arm | No Pretreatment Arm
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No